CLINICAL TRIAL: NCT03603938
Title: Effect of Potassium Losartan With Bedtime Dosing on Chronic Kidney Disease Patients With Nondipping Blood Pressure Pattern
Brief Title: Bedtime Potassium Losartan on CKD With Nocturnal Hypertension Patients With Nondipping Blood Pressure Pattern
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cheng Wang, Director of Nephrology Department, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.SNK.002
Record Dates: First submitted 2018-07-04; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Chronic Kidney Disease Patients
Keywords: potassium losartan, CKD, nondipping BP pattern
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bedtime dosing ARB for hypertension (Experimental): potassium losartan has benefit for the nondipping BP pattern
  Interventions: Drug: potassium losartan
- bedtime dosing ARB for the prognosis (Experimental): bedtime administration of potassium losartan has benefit for the prognosis of CKD patients
  Interventions: Drug: potassium losartan

INTERVENTIONS:
Drug: potassium losartan — treated with bedtime or awakening doses of potassium losartan
  Other Names: Kesiya

SUMMARY:
Nondipping blood pressure (BP) pattern is a potential independent risk factor for chronic kidney disease (CKD). Whether bedtime administration of potassium losartan has benefit for anti-hypertension and the prognosis of CKD patients is not clear. Patients with nondipping BP pattern or dipping BP pattern were enrolled in this study, and the patients with nondipping BP pattern were randomly divided into two groups and treated with bedtime or awakening doses of potassium losartan.

DETAILED DESCRIPTION:
Patients with nondipping BP pattern or dipping BP pattern were enrolled in this study, and the patients with nondipping BP pattern were randomly divided into two groups and treated with bedtime or awakening doses of potassium losartan. Any patients who had any antihypertension medication at bedtime would withdrawal the drugs for 2 weeks before ABPM. Patients with nondipping BP were then randomly divided into two groups and received a bedtime or awakening dose of potassium losartan. Patients with dipping BP were called the dipper group, while the patients with nondipping BP were called the awakening dose group or bedtime dose group, according to the time of drug administration.

ELIGIBILITY:
Inclusion Criteria:

* night BP is SBP≥120mmHg and/or DBP≥70mmHg；
* presence of CKD;
* estimated GFR (eGFR)<90 mL⁄ min ⁄ 1.73 m2 (using the Modification of Diet in Renal Disease Study equation) but >30 mL⁄ min ⁄1.73 m2;
* signed informed consent from participating patients.

Exclusion Criteria:

* pregnancy;
* tumor;
* infection;
* renal replacement;
* history of drug or alcohol abuse;
* night- or shift-work employment;
* treatment with steroids or hormonal therapy;
* acute changes in eGFR >30% in the past 3 months;
* presence of acquired immunodeficiency syndrome;
* CV disorders (unstable angina pectoris, heart failure, life-threatening arrhythmia, atrial fibrillation, kidney failure,and grade III or IV retinopathy);
* intolerance to ambulatory BP monitoring (ABPM);
* inability to communicate and comply with all of the study requirements.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
renal events and Cardiovascular events | 5 years
  doubled creatine or renal replacement, myocardial infarction, heart failure, stroke, vascular reconstruction, peripheral vascular disease, non-traumatic amputation

SECONDARY OUTCOMES:
proteinuria | 5 years
  24h proteinuria >1g
renal function | 5 years
  eGFR<30ml/min/1.73m2
Thickness of the medial membrane of the carotid artery | 5 years
  cIMT >1mm
Left ventricle weight index | 5 years
  LVMI >115g/m2 (man) 和 >95g/m2 (woman)

CONTACTS AND LOCATIONS:
Overall Officials: Shaoxuan Liu, Study Chair — GCP Office
Locations (1):
- The fifth affiliated hospital of Sun Yat-sen university, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Liu ZH. Nephrology in china. Nat Rev Nephrol. 2013 Sep;9(9):523-8. doi: 10.1038/nrneph.2013.146. Epub 2013 Jul 23. PMID 23877587
- [Background] Zheng Y, Cai GY, Chen XM, Fu P, Chen JH, Ding XQ, Yu XQ, Lin HL, Liu J, Xie RJ, Wang LN, Ni ZH, Liu FY, Yin AP, Xing CY, Wang L, Shi W, Liu JS, He YN, Ding GH, Li WG, Wu GL, Miao LN, Chen N, Su Z, Mei CL, Zhao JY, Gu Y, Bai YK, Luo HM, Lin S, Chen MH, Gong L, Yang YB, Yang XP, Li Y, Wan JX, Wang NS, Li HY, Xi CS, Hao L, Xu Y, Fang JA, Liu BC, Li RS, Wang R, Zhang JH, Wang JQ, Lou TQ, Shao FM, Mei F, Liu ZH, Yuan WJ, Sun SR, Zhang L, Zhou CH, Chen QK, Jia SL, Gong ZF, Guan GJ, Xia T, Zhong LB; Prevalence, Awareness, and Treatment Rates in Chronic Kidney Disease Patients with Hypertension in China (PATRIOTIC) Collaborative Group. Prevalence, awareness, treatment, and control of hypertension in the non-dialysis chronic kidney disease patients. Chin Med J (Engl). 2013 Jun;126(12):2276-80. PMID 23786938
- [Background] Luan FL, Norman SP. Intensive blood-pressure control in hypertensive chronic kidney disease. N Engl J Med. 2010 Dec 23;363(26):2564-5; author reply 2565-6. doi: 10.1056/NEJMc1011419. No abstract available. PMID 21175325
- [Background] Hodgkinson J, Mant J, Martin U, Guo B, Hobbs FD, Deeks JJ, Heneghan C, Roberts N, McManus RJ. Relative effectiveness of clinic and home blood pressure monitoring compared with ambulatory blood pressure monitoring in diagnosis of hypertension: systematic review. BMJ. 2011 Jun 24;342:d3621. doi: 10.1136/bmj.d3621. PMID 21705406
- [Background] Lv J, Ehteshami P, Sarnak MJ, Tighiouart H, Jun M, Ninomiya T, Foote C, Rodgers A, Zhang H, Wang H, Strippoli GF, Perkovic V. Effects of intensive blood pressure lowering on the progression of chronic kidney disease: a systematic review and meta-analysis. CMAJ. 2013 Aug 6;185(11):949-57. doi: 10.1503/cmaj.121468. Epub 2013 Jun 24. PMID 23798459
- [Background] Fan HQ, Li Y, Thijs L, Hansen TW, Boggia J, Kikuya M, Bjorklund-Bodegard K, Richart T, Ohkubo T, Jeppesen J, Torp-Pedersen C, Dolan E, Kuznetsova T, Stolarz-Skrzypek K, Tikhonoff V, Malyutina S, Casiglia E, Nikitin Y, Lind L, Sandoya E, Kawecka-Jaszcz K, Imai Y, Ibsen H, O'Brien E, Wang J, Staessen JA; International Database on Ambulatory Blood Pressure In Relation to Cardiovascular Outcomes Investigators. Prognostic value of isolated nocturnal hypertension on ambulatory measurement in 8711 individuals from 10 populations. J Hypertens. 2010 Oct;28(10):2036-45. doi: 10.1097/HJH.0b013e32833b49fe. PMID 20520575
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] O'Brien E, Sheridan J, O'Malley K. Dippers and non-dippers. Lancet. 1988 Aug 13;2(8607):397. doi: 10.1016/s0140-6736(88)92867-x. No abstract available. PMID 2899801
- [Background] Iimuro S, Imai E, Watanabe T, Nitta K, Akizawa T, Matsuo S, Makino H, Ohashi Y, Hishida A; Chronic Kidney Disease Japan Cohort Study Group. Clinical correlates of ambulatory BP monitoring among patients with CKD. Clin J Am Soc Nephrol. 2013 May;8(5):721-30. doi: 10.2215/CJN.06470612. Epub 2013 Feb 14. PMID 23411432
- [Background] Hering D. Predictive Role of Nighttime Blood Pressure in Response to Renal Denervation: Evidence From the DENER-HTN Study (Renal Denervation for Hypertension). Hypertension. 2017 Mar;69(3):398-400. doi: 10.1161/HYPERTENSIONAHA.116.08738. Epub 2017 Jan 23. No abstract available. PMID 28115511
- [Background] Hansen TW, Li Y, Boggia J, Thijs L, Richart T, Staessen JA. Predictive role of the nighttime blood pressure. Hypertension. 2011 Jan;57(1):3-10. doi: 10.1161/HYPERTENSIONAHA.109.133900. Epub 2010 Nov 15. PMID 21079049
- [Background] Yano Y, Kario K. Nocturnal blood pressure and cardiovascular disease: a review of recent advances. Hypertens Res. 2012 Jul;35(7):695-701. doi: 10.1038/hr.2012.26. Epub 2012 Mar 1. PMID 22378470
- [Background] Li Y, Staessen JA, Lu L, Li LH, Wang GL, Wang JG. Is isolated nocturnal hypertension a novel clinical entity? Findings from a Chinese population study. Hypertension. 2007 Aug;50(2):333-9. doi: 10.1161/HYPERTENSIONAHA.107.087767. Epub 2007 Jun 18. PMID 17576859
- [Background] Sarnak MJ, Levey AS, Schoolwerth AC, Coresh J, Culleton B, Hamm LL, McCullough PA, Kasiske BL, Kelepouris E, Klag MJ, Parfrey P, Pfeffer M, Raij L, Spinosa DJ, Wilson PW; American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Kidney disease as a risk factor for development of cardiovascular disease: a statement from the American Heart Association Councils on Kidney in Cardiovascular Disease, High Blood Pressure Research, Clinical Cardiology, and Epidemiology and Prevention. Hypertension. 2003 Nov;42(5):1050-65. doi: 10.1161/01.HYP.0000102971.85504.7c. No abstract available. PMID 14604997
- [Background] Pogue V, Rahman M, Lipkowitz M, Toto R, Miller E, Faulkner M, Rostand S, Hiremath L, Sika M, Kendrick C, Hu B, Greene T, Appel L, Phillips RA; African American Study of Kidney Disease and Hypertension Collaborative Research Group. Disparate estimates of hypertension control from ambulatory and clinic blood pressure measurements in hypertensive kidney disease. Hypertension. 2009 Jan;53(1):20-7. doi: 10.1161/HYPERTENSIONAHA.108.115154. Epub 2008 Dec 1. PMID 19047584
- [Background] Perez-Lloret S, Toblli JE, Cardinali DP, Malateste JC, Milei J. Nocturnal hypertension defined by fixed cut-off limits is a better predictor of left ventricular hypertrophy than non-dipping. Int J Cardiol. 2008 Jul 21;127(3):387-9. doi: 10.1016/j.ijcard.2007.04.027. Epub 2007 Jun 15. PMID 17574691
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Bedtime dosing of antihypertensive medications reduces cardiovascular risk in CKD. J Am Soc Nephrol. 2011 Dec;22(12):2313-21. doi: 10.1681/ASN.2011040361. Epub 2011 Oct 24. PMID 22025630
- [Background] Rahman M, Greene T, Phillips RA, Agodoa LY, Bakris GL, Charleston J, Contreras G, Gabbai F, Hiremath L, Jamerson K, Kendrick C, Kusek JW, Lash JP, Lea J, Miller ER 3rd, Rostand S, Toto R, Wang X, Wright JT Jr, Appel LJ. A trial of 2 strategies to reduce nocturnal blood pressure in blacks with chronic kidney disease. Hypertension. 2013 Jan;61(1):82-8. doi: 10.1161/HYPERTENSIONAHA.112.200477. Epub 2012 Nov 19. PMID 23172931
- [Background] Verdecchia P, Angeli F, Mazzotta G, Garofoli M, Ramundo E, Gentile G, Ambrosio G, Reboldi G. Day-night dip and early-morning surge in blood pressure in hypertension: prognostic implications. Hypertension. 2012 Jul;60(1):34-42. doi: 10.1161/HYPERTENSIONAHA.112.191858. Epub 2012 May 14. PMID 22585951
- [Background] Schillaci G, Battista F, Settimi L, Schillaci L, Pucci G. Antihypertensive drug treatment and circadian blood pressure rhythm: a review of the role of chronotherapy in hypertension. Curr Pharm Des. 2015;21(6):756-72. doi: 10.2174/1381612820666141024130013. PMID 25341857
- [Background] Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol. 2002 Jul 1;90(1):29-34. doi: 10.1016/s0002-9149(02)02381-0. PMID 12088775
- [Background] Dudeja SK, Dudeja RK. Blood-pressure measurement. N Engl J Med. 2009 May 7;360(19):2034-5; author reply 2035. No abstract available. PMID 19425241
- [Result] Wang C, Zhang J, Liu X, Li CC, Ye ZC, Peng H, Chen Z, Lou T. Effect of valsartan with bedtime dosing on chronic kidney disease patients with nondipping blood pressure pattern. J Clin Hypertens (Greenwich). 2013 Jan;15(1):48-54. doi: 10.1111/jch.12021. Epub 2012 Oct 9. PMID 23282124
- [Result] Wang C, Li Y, Zhang J, Ye Z, Zhang Q, Ma X, Peng H, Lou T. Prognostic Effect of Isolated Nocturnal Hypertension in Chinese Patients With Nondialysis Chronic Kidney Disease. J Am Heart Assoc. 2016 Oct 10;5(10):e004198. doi: 10.1161/JAHA.116.004198. PMID 27792646
- [Result] Wang C, Deng WJ, Gong WY, Zhang J, Tang H, Peng H, Zhang QZ, Ye ZC, Lou T. High prevalence of isolated nocturnal hypertension in Chinese patients with chronic kidney disease. J Am Heart Assoc. 2015 Jun 18;4(6):e002025. doi: 10.1161/JAHA.115.002025. PMID 26089178
- [Result] Wang C, Deng WJ, Gong WY, Zhang J, Zhang QZ, Ye ZC, Lou T. Nocturnal Hypertension Correlates Better With Target Organ Damage in Patients With Chronic Kidney Disease than a Nondipping Pattern. J Clin Hypertens (Greenwich). 2015 Oct;17(10):792-801. doi: 10.1111/jch.12589. Epub 2015 Jun 4. PMID 26041362